CLINICAL TRIAL: NCT03180229
Title: Granisetron Effect on Hemodynamic Changes and Intubation Condition During Anesthesia Induction in Laparoscopic Cholecystectomy
Brief Title: Granisetron Effect on Hemodynamic Changes in Laparoscopic Cholecystectomy
Acronym: lap
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Diskapi
Record Dates: First submitted 2017-05-29; First posted 2017-06-08 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Granisetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granisetron (Active Comparator): Five minutes before the induction 1 ml (1 mg / ml) iv granisetron will use. .Then blood pressure (systolic, diastolic, mean) and heart rate will record per 5 minute during surgery.
  Interventions: Drug: Granisetron 1 Mg/mL Intravenous Solution
- Control (No Intervention): Five minutes before the induction 1 ml saline iv use.Then blood pressure (systolic, diastolic, mean) and heart rate will record per 5 minute during surgery.

INTERVENTIONS:
Drug: Granisetron 1 Mg/mL Intravenous Solution — 1 milligram (mg) will use on group Granisetron before 5 min induction
  Arms: Granisetron

SUMMARY:
Propofol is one of the most commonly used anesthetic agents because of its ability to induce rapid and reliable collection. However, hypotension and injection pain in the induction are the most common complications. After induction of propofol; The cardiovascular system depresses, resulting in a drop in blood pressure due to decreased cardiac output and systemic vascular resistance. This may also contribute to the reduction of sympathetic tone activity in the central way, and slight reduction in the number of pulses that develop as a result of increasing vagal activity. İn order to attenuate these hemodynamic undesired effects caused by propofol, various agents were tried such as atropine, ephedrine, volume replacement ringer lactate, ketamine. Ondansetron and granisetron, which are used for postoperative nausea and vomiting prophylaxis, have been used as such. Therefore, ondansetron and granisetron were preventing hypotension induced by post-spinal and general anesthesia induction.

The investigator also tried to demonstrate the effect of granisetron, another serotonin type 3 (5-HT3) receptor antagonist for postoperative nausea and vomiting prophylaxis, on induction hypotension and intubation quality after propofol induction in this study

DETAILED DESCRIPTION:
150 participants with American Society of Anesthesiologists (ASA) physical score I-II who underwent elective laparoscopic cholecystectomy between the ages of 18-70 will be enrolled. Participants will be divided into two groups using granisetron and control.

All participants will be premedicated with 0.05 mg kg-1 midazolam 30 minutes before the operation. ASA, age, sex, weight demographic data of the participants who were taken to the operating room will record. Peripheral oxygen saturation (SPO2), noninvasive blood pressure and electrocardiography (ECG) will monitored. A venous cannula will place on the back of the hand. Participants will randomly divide into 2 groups by closed envelope method.

Five minutes before the induction of group G, 1 ml (1 mg / ml) iv granisetron, group K will receive 1 ml saline. Propofol at induction will be administered at a dose of 0.6 mg / kg of rocuronium at a dose of 2 mg / kg. Pre-induction, post-intubation and every five minutes SPO2, diastolic arterial pressure (DAP), mean arterial pressure (MAP), systolic arterial pressure(SAP) and heart rate (HR) will record. Intubation quality will be evaluated by evans score.

Systolic Blood Pressure <Control + 15 0 <Control + 30 1 1

* Control + 30 2 Heart Rate Pressure <Control + 15 0 <Control + 30 1
* Control + 30 2 Sweating No 0 Moist leather 1 Visible sweating 2 Tears No 0 Yes 1 Overflowing 2

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic Cholecystectomy (lap) surgery

Exclusion Criteria:

* Acute pancreatitis disease
* Cardiorespiratory disease
* Hypertension
* Anti hypertension treatments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-70
Enrollment: 140 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
change mean arterial blood pressure | Change from Baseline Systolic Blood Pressure at per 5 minute during surgery
  mean arterial blood pressure (MAP) MAP at least 25% less than the basal value
intubation quality | intubation period
  in this time evans score which is included tears, sweating, systolic arterial blood pressure and heart rate will be used. the change baseline systolic arterial blood pressure and heart rate and tears, sweating will score numeric.
change heart rate | Change from baseline heart rate at per 5 minute during surgery
  HR <60 or >25% drop baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital Ankara, Turkey, Ankara, Turkey (Türkiye)